CLINICAL TRIAL: NCT03886922
Title: The Hemodynamics Effect of Levcromakalim After Glibenclamide Administration Assessed by High Resolution MRA Technique in a Randomized, Double-blind, Cross-over and Placebo-controlled Study With Healthy Volunteers.
Brief Title: The Hemodynamics Effect of Glibenclamide on Levcromakalim Assessed by High Resolution Magnetic Resonance Angiography (MRA) Technique in a Randomized Double-blind Cross-over Placebo-controlled Study With Healthy Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Mohammad Al-Mahdi Al-Karagholi, MD, PhD student, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: Glibenclamide H-18052188
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Hemodynamics of Cranial Arteries; Headache; Cerebral Blood Flow
MeSH Terms: conditions — Headache | interventions — Cromakalim; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, cross-over, placebo-controlled design in healthy volunteers.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Glibenclamide and Levcromakalim (Active Comparator): Participants will receive levcromakalim infusion after glibenclamide administration
  Interventions: Drug: Levcromakalim
- Glibenclamide and Saline (Active Comparator): Participants will receive placebo infusion after glibenclamide administration
  Interventions: Drug: Saline
- Placebo (Sham Comparator): Participants will receive placebo infusion after placebo administration.
  Interventions: Drug: Saline
- Levcromakalim and Glibenclamide (Active Comparator): Participants will receive levcromakalim infusion before glibenclamide administration.
  Interventions: Drug: Levcromakalim
- Levcromakalim and Placebo (Active Comparator): Participants will receive levcromakalim infusion before placebo administration.
  Interventions: Drug: Levcromakalim; Drug: Saline

INTERVENTIONS:
Drug: Levcromakalim — Intravenous infusion of levcromakalim or placebo for 20 minutes. To investigate the role of levcromakalim/placebo on cranial arteries in healthy volunteers after glibenclamide administration.
  Arms: Glibenclamide and Levcromakalim; Levcromakalim and Glibenclamide; Levcromakalim and Placebo
Drug: Saline — Intravenous infusion of levcromakalim or placebo for 20 minutes. To investigate the role of levcromakalim/placebo on cranial arteries in healthy volunteers after glibenclamide administration.
  Arms: Glibenclamide and Saline; Levcromakalim and Placebo; Placebo

SUMMARY:
To investigate the effect of levcromakalim/placebo infusion on cranial arteries after glibenclamide administration.

DETAILED DESCRIPTION:
15 healthy participants will randomly be allocated to receive levcromakalim or placebo on to different days before and after oral glibenclamide administration.

The aim of the study is to investigate the effect of levcromakalim/placebo infusion on cranial arteries before and after glibenclamide administration.

Repeated magnetic resonance angiography (MRA) measurements covering the middle meningeal artery (MMA), superficial temporal artery (STA) and middle cerebral artery (MCA) before and after glibenclamide administration and levcromakalim/placebo infusion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both sexes.
* 18-60 years.
* 50-100 kg.
* Women of childbearing potential must use adequate contraception

Exclusion Criteria:

* A history of serious somatic disease
* Migraine or any other type of headache (except episodic tension-type headache less than once a month)
* Daily intake of any medication except contraceptives
* Contraindications for MRI scan.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the middle meningeal artery (MMA), superficiel temporal artery (STA) and middle cerebral artery (MCA) | Time of measurements is baseline, 1 hour after glibenclamide administration, 2 hour after glibenclamide administration, 20 minutes after levcromakalim infusion, 60 min after levcromakalim infusion
  Repeated MRA measurements covering the diameter of MMA , STA and MCA before and after glibenclamide administration and levcromakalim/placebo infusion measured by centimeter (cm)
Changes in Cerebral blood flow | Time of measurements is baseline, 1 hour after glibenclamide administration, 2 hour after glibenclamide administration, 20 minutes after levcromakalim infusion, 60 min after levcromakalim infusion
  Repeated MRA measurements covering the blood flow before and after glibenclamide administration and levcromakalim/placebo infusion measured by centimeter (cm)/minutes
Headache | Time of headache measurements is from before (-10 min) and after (12 hours) glibenclamide administration.
  Headache intensity will be recorded by numerical rating scale (NRS) from 0 to 10 (0, no headache; 1, a feeling of pressure; 10, worst imaginable headache).

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Danish headache center, Glostrup Municipality, Copenhagen
  - Mohammad Al-Mahdi Al-Karagholi, København S, Danmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Al-Karagholi MA, Ghanizada H, Kokoti L, Paulsen JS, Hansen JM, Ashina M. Effect of KATP channel blocker glibenclamide on levcromakalim-induced headache. Cephalalgia. 2020 Sep;40(10):1045-1054. doi: 10.1177/0333102420949863. Epub 2020 Aug 17. PMID 32806954